CLINICAL TRIAL: NCT03777423
Title: Evaluation of Biting Force of Removable Partial Denture Made of Injection Molded PEEK Framework Versus Cobalt Chromium Framework in Mandibular Kennedy Class I Edentulous Cases
Brief Title: Comparison Between Injection Molded PEEK Framework and Cobalt Chromium Framework Removable Partial Dentures Regarding Biting Force
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Hatim Mohammed, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-11-29
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Mandibular Prosthesis User

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK framework partial dentures (Experimental): High performance ketone polymers introduced lately.These polymer-based frameworks provide better esthetics, higher elasticity, lighter in weight, have low water sorption and solubility, and are easily repaired and reproduced.
  Interventions: Device: PEEK framework partial dentures
- Cobalt-chromium framework partial dentures (Active Comparator): it is considered the gold standard framework. These frameworks are less bulky with high strength, conduct heat and electricity well, and have good durability. some disadvantages include hypersensitivity, adverse tissue reactions and bad aesthetics.
  Interventions: Device: Cobalt- chromium framework partial dentures

INTERVENTIONS:
Device: PEEK framework partial dentures — Polymer-based framework recently introduced made of polyetheretherketone polymer frame combined with acrylic resin denture teeth and a conventional acrylic resin denture base.
  Arms: PEEK framework partial dentures
Device: Cobalt- chromium framework partial dentures — It's a bio-compatible metal used in thin sections so less bulky, provide high strength and stiffness ,conduct heat and cold for a more natural experience, enable designs that minimize the covering of the gingival margins, allow for a stable denture base, and resistance to corrosion.Drawbacks of metal frameworks can include hypersensitivity, aesthetics because of metal metal display, oral galvanism, adverse tissue reactions, osteolysis of abutment teeth, and biofilm production
  Arms: Cobalt-chromium framework partial dentures

SUMMARY:
This study is aiming to evaluate the biting force of polyetheretherketone (PEEK) framework partial dentures compared to that of cobalt-chromium ones in mandibular Kennedy class I edentulous cases hoping that polyetheretherketone (PEEK) framework removable partial dentures can improve the patient masticatory efficiency .

ELIGIBILITY:
Inclusion Criteria:

-Kennedy class 1 partially edentulous subjects indicated for framework partial denture

Exclusion Criteria:

* Uncooperative patients
* Bad oral hygiene patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Biting force | Change in baseline biting force from time of insertion, insertion after 1 month and after 3 months
  Biting force of the patient wearing the removable partial denture measured by I-load sensor device.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of oral and dental medincine Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Al-Jammali ZM. Clinical Evaluation of Maximum Bite Force in Patient with Heat Cure acrylic and Flexible Partial Dentures. Medical Journal of Babylon. 2017;14(3):509-17.